CLINICAL TRIAL: NCT04116632
Title: A Multiple Dose Pharmacokinetic/Pharmacodynamic and Safety and Tolerability Study of BMS-963272 in Obese But Otherwise Healthy Adults
Brief Title: A Multiple Dose Study to Assess the Safety and Tolerability of BMS-963272 in Obese But Otherwise Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB006-017
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Obese But Otherwise Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-963272 or Placebo once daily (QD) (Experimental)
  Interventions: Drug: BMS-963272; Drug: Placebo
- BMS-963272 or Placebo every 12 hours (Q12H) (Experimental)
  Interventions: Drug: BMS-963272; Drug: Placebo
- BMS-963272 or Placebo every 8 hours (Q8H) (Experimental)
  Interventions: Drug: BMS-963272; Drug: Placebo

INTERVENTIONS:
Drug: BMS-963272 — Single dose with varying frequency among groups
Drug: Placebo — Specified dose on specified days

SUMMARY:
This study will assess the safety and tolerability of multiple doses of BMS-963272 in obese but otherwise healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants must be in good general health, in the opinion of the investigator, with no clinically significant deviation from normal in medical history, physical examination findings, ECGs, or laboratory results.
* Participants must have a BMI of 30 kg/m2 to 40 kg/m2 inclusive
* Women (not of childbearing potential) and men aged 18 to 60 years, inclusive

Exclusion Criteria:

* Previous participation in the current study
* Inability or unwillingness to comply with protocol-defined restrictions or requirements regarding lifestyle, diet, concomitant medications, or other aspects of the study
* Inability to tolerate the oLTT meal or to comply with oLTT testing conditions
* Inability to tolerate oral medication
* Inability to tolerate venipuncture and/or inadequate venous access
* Women who are breastfeeding
* Medical Conditions
* History of lactose intolerance
* Any significant (in the opinion of the investigator) acute or chronic illness
* Type 1 or 2 diabetes
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population
* Previous/Concomitant Therapy
* Previous exposure to BMS-963272

Other protocol-defined inclusion/exclusion criteria could apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of BMS-963272 (Cmax) | Day 1, Day 14
Time of maximum observed concentration of BMS-963272 (Tmax) | Day 1, Day 14
Area under the concentration-time curve in one dosing interval (AUC(TAU)) | Day 1, Day 14
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) | Day 14
Apparent total clearance of the drug from plasma after oral administration (CLss/F) | Day 14
Apparent volume of distribution at steady state (Vss/F) | Day 14
Average concentration at steady state (Cavg,ss) | Day 14
Half-life (T-HALF) | Day 14
Accumulation index (AI) | Day 14
Rate elimination constant (kel) of BMS-963272 | Day 14
Area under the concentration-time curve (AUC) of triglycerides (TG) and fatty acids in response to the oral lipid tolerance test (oLTT) | Day 7, Day 15
Incremental AUC (iAUC) of TG and fatty acids in response to the oLTT | Day 7, Day 15

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 55 days
Incidence of Serious Adverse Events (SAEs) | Up to 55 days
Number of clinically significant changes in vital signs, electrocardiograms (ECGs), physical examinations and clinical laboratory tests | Up to 55 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Lenexa, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm